CLINICAL TRIAL: NCT02499289
Title: Does Prolonged Fasting Break the Vicious Circle of Polycystic Ovarian Syndrome of Insulin Resistance ?
Brief Title: Effect of Ramadan Fasting on Ovulation and Insuline Resistance in Patients With PCOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, Dr. Ahmed Kotb, Ain Shams University
Other Study IDs: PCOS FASTING
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Polycystic ovary syndrome (PCOS) has a heterogeneous clinical presentation comprising reproductive (hyperandrogenism, menstrual irregularity, anovulation, infertility, pregnancy complications), metabolic [insulin resistance (IR), increased type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD) risk factors] and psychological features (worsened quality of life and increased anxiety and depression) Whether prolonged fasting during Ramadan breaks the insulin resistance state of polycystic ovarian syndrome and subsequently improve the ovulation and spontaneous pregnancy will happen without ovarian stimulation.

DETAILED DESCRIPTION:
Question of the study:

The question is raised whether prolonged fasting during Ramadan breaks the insulin resistance state of polycystic ovarian syndrome and improve the metabolic syndrome does prolonged fasting decrease glucose level, insulin level, insulin resistance markers such as adipokines and subsequently improve ovarian function and causes spontaneous ovulation.

ELIGIBILITY:
Inclusion Criteria:

* Females with PCO in child bearing age who presented at reproductive and endocrinology clinics at Ain Shams University Maternity Hospital, and welling to fast for 30 days from 5 am until 7 pm and do not plan to induce her ovulation in the next 4 months to get pregnant.
* Does not have any other medical illnesses other than PCO.
* Welling not to start any ovulation induction in the next 4 months after the first blood sample was taken and after fasting month.

Exclusion Criteria:

* Known androgen secreting tumor.
* PCO on ovarian stimulation medications
* PCO with any other medical illness.
* Non-compliance with fasting 30 days from 5 am- 7 pm.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: • Females with PCO in child bearing age who presented at reproductive and endocrinology clinics at Ain Shams University Maternity Hospital, and welling to fast for 30 days from 5 am until 7 pm and do not plan to induce her ovulation in the next 4 months to get pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
spontaneous ovulation measured by midluteal progesterone | one month
  Ovulation will be monitored by the Progesterone level on 22nd day of first cycle after 30 days of prolonged daily Fasting (Ramadan).

SECONDARY OUTCOMES:
clinical pregnancy | four months
  We will record any pregnancy will happened in the next 4 months after Fasting without any ovulation induction.
fasting glucose/insuline ratio | one month
  Insulin resistance (IR) measuring: fasting 8 hours. Plasma glucose (FPG) and fasting insulin (FIN) will be measured by chemiluminescent immunoassay. The ratio of glucose/insulin represents the degree of IR
Plasma adiponectin | one month
  Plasma adiponectin will be measured before and after 30 days fasting
plasma resistin | one month
  Plasma resistin will be measured before and after 30 days fasting
plasma gherlin | one month
  Plasma gherlin will be measured before and after 30 days fasting

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided